CLINICAL TRIAL: NCT02554682
Title: A Pilot Efficacy and Implementation Study of the Patients, Parents and Professionals Partnering to Improve Adolescent Health (P4) Intervention
Brief Title: The P4 Intervention Study to Improve Adolescent Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 15-011732
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Adolescent Behavior
Keywords: Adolescent Health; Sexual Health; Parent-Teen Communication; Teen Driving; Alcohol Prevention
MeSH Terms: conditions — Adolescent Behavior | interventions — Sexual Health; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sexual Health (Other): Parents of teens between the ages of 14 and 15 will review psychoeducational workbooks related to sexual health at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Interventions: Behavioral: Sexual Health
- Alcohol Prevention (Other): Parents of teens between the ages of 14 and 15 will review psychoeducational workbooks related to alcohol prevention at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Interventions: Behavioral: Alcohol Prevention
- Sexual Health & Alcohol Control Group (No Intervention): Parents of teens between the ages of 14 and 15 will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 4 to 5 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from both the sexual health and alcohol prevention groups.
- Teen Driving (Other): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will review psychoeducational workbooks related to teen driving at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 6 months post baseline we will collect data to assess the effectiveness of the study materials.
  Interventions: Behavioral: Teen Driving
- Teen Driving Control (No Intervention): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.

INTERVENTIONS:
Behavioral: Sexual Health — Psychoeducational workbook, worksheets, tip sheets, and health coaching session about sexual health, sexually transmitted disease (STD) prevention, and safe sex practices for teenager.
  Arms: Sexual Health
Behavioral: Alcohol Prevention — Psychoeducational workbook, worksheets, tip sheets, and health coaching session about alcohol prevention and safety, underage drinking, and drinking and driving.
  Arms: Alcohol Prevention
Behavioral: Teen Driving — Psychoeducational workbook, worksheets, videos, tip sheets, and health coaching session about how parents can help supervise their teens' safe driving practices and how to talk with their teen about important safety topics for teen drivers.
  Arms: Teen Driving

SUMMARY:
The primary objective is to conduct a pilot study to determine the efficacy of evidence-based interventions delivered in primary care clinic settings on parent-teen health communication.

DETAILED DESCRIPTION:
Primary care provides a means by which to connect evidence-based interventions with patients; however, many interventions have been evaluated using randomized controlled trials (RCTs) in non-healthcare settings.

The primary objective is to conduct a pilot study to determine the effect of evidence-based interventions delivered in primary care clinic settings on parent-teen communication about alcohol use, sexual health, and safe driving.

Eligible participants are healthy adolescent patients from the Children's Hospital of Philadelphia (CHOP) primary care network with a well-child visit scheduled between the ages of 14 to 17 years with one parent willing to participate. Adolescents that hold an intermediate driver's license, that are pregnant, or that have pervasive development disorder or a developmental delay are excluded from this study.

Parents will be given written psychoeducational intervention materials on communicating with their adolescents about alcohol use, sexual health, or safe driving (e.g.,booklets, tip sheet brochures, activity workbooks, web links), receive coaching about using the intervention materials, and provider endorsement of the materials during the well-child visit, as well as follow-up phone health coaching 2 weeks after the appointment.

The primary endpoints are evaluating the difference between the intervention and control groups on parent-teen communication on the targeted health topics.

ELIGIBILITY:
Inclusion Criteria:

1. CHOP Primary Care patient
2. Scheduled for a well-child visit that parent and teen both plan to attend within 3 weeks of enrollment
3. [Teen Driving Arm Only] Planning on having the medical certification for the permit application completed at their next well child visit and planning on taking their driving permit test in the next 8 weeks

Exclusion Criteria:

1. Not fluent in written or spoken English
2. Developmental Delay or Pervasive Developmental Disorder
3. Pregnant female
4. [Teen Driving Arm Only] Already has driving permit (has taken and passed the knowledge test) and/or the medical certification for the permit application was not completed at the well child visit

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Ford, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kann L, Kinchen S, Shanklin SL, Flint KH, Kawkins J, Harris WA, Lowry R, Olsen EO, McManus T, Chyen D, Whittle L, Taylor E, Demissie Z, Brener N, Thornton J, Moore J, Zaza S; Centers for Disease Control and Prevention (CDC). Youth risk behavior surveillance--United States, 2013. MMWR Suppl. 2014 Jun 13;63(4):1-168. PMID 24918634
- [Background] Sales JM, Milhausen RR, Wingood GM, Diclemente RJ, Salazar LF, Crosby RA. Validation of a Parent-Adolescent Communication Scale for use in STD/HIV prevention interventions. Health Educ Behav. 2008 Jun;35(3):332-45. doi: 10.1177/1090198106293524. Epub 2006 Dec 15. PMID 17200099
- [Background] Ford CA, Cheek C, Culhane J, Fishman J, Mathew L, Salek EC, Webb D, Jaccard J. Parent and Adolescent Interest in Receiving Adolescent Health Communication Information From Primary Care Clinicians. J Adolesc Health. 2016 Aug;59(2):154-61. doi: 10.1016/j.jadohealth.2016.03.001. Epub 2016 Apr 14. PMID 27151760
- [Background] Ford CA, Davenport AF, Meier A, McRee AL. Partnerships between parents and health care professionals to improve adolescent health. J Adolesc Health. 2011 Jul;49(1):53-7. doi: 10.1016/j.jadohealth.2010.10.004. Epub 2011 Mar 12. PMID 21700157
- [Background] Guilamo-Ramos V, Jaccard J, Turrisi R, Johansson M. Parental and school correlates of binge drinking among middle school students. Am J Public Health. 2005 May;95(5):894-9. doi: 10.2105/AJPH.2003.018952. PMID 15855471
- [Background] Guilamo-Ramos V, Bouris A, Jaccard J, Gonzalez B, McCoy W, Aranda D. A parent-based intervention to reduce sexual risk behavior in early adolescence: building alliances between physicians, social workers, and parents. J Adolesc Health. 2011 Feb;48(2):159-63. doi: 10.1016/j.jadohealth.2010.06.007. PMID 21257114
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2009. Natl Vital Stat Rep. 2010 Dec;59(3):1-19. PMID 25073731
- [Background] Jaccard J, Dodge T, Dittus P. Parent-adolescent communication about sex and birth control: a conceptual framework. New Dir Child Adolesc Dev. 2002 Fall;(97):9-41. doi: 10.1002/cd.48. No abstract available. PMID 14964942
- [Background] Kerr M, Stattin H. What parents know, how they know it, and several forms of adolescent adjustment: further support for a reinterpretation of monitoring. Dev Psychol. 2000 May;36(3):366-80. PMID 10830980
- [Background] Mayhew DR, Simpson HM, Pak A. Changes in collision rates among novice drivers during the first months of driving. Accid Anal Prev. 2003 Sep;35(5):683-91. doi: 10.1016/s0001-4575(02)00047-7. PMID 12850069
- [Background] McCartt AT, Shabanova VI, Leaf WA. Driving experience, crashes and traffic citations of teenage beginning drivers. Accid Anal Prev. 2003 May;35(3):311-20. doi: 10.1016/s0001-4575(02)00006-4. PMID 12643948
- [Background] Mirman JH, Curry AE, Winston FK, Wang W, Elliott MR, Schultheis MT, Fisher Thiel MC, Durbin DR. Effect of the teen driving plan on the driving performance of teenagers before licensure: a randomized clinical trial. JAMA Pediatr. 2014 Aug;168(8):764-71. doi: 10.1001/jamapediatrics.2014.252. PMID 24957844
- [Background] Mirman JH, Albert WD, Curry AE, Winston FK, Fisher Thiel MC, Durbin DR. TeenDrivingPlan effectiveness: the effect of quantity and diversity of supervised practice on teens' driving performance. J Adolesc Health. 2014 Nov;55(5):620-6. doi: 10.1016/j.jadohealth.2014.04.010. Epub 2014 Jun 9. PMID 24925492
- [Background] Olson, D. H.. Family inventories: Inventories used in a national survey of families across the life cycle. St Paul, MN: Family Social Science, University of Minnesota. 1985
- [Background] Stattin H, Kerr M. Parental monitoring: a reinterpretation. Child Dev. 2000 Jul-Aug;71(4):1072-85. doi: 10.1111/1467-8624.00210. PMID 11016567
- [Background] Turrisi R, Jaccard J, Taki R, Dunnam H, Grimes J. Examination of the short-term efficacy of a parent intervention to reduce college student drinking tendencies. Psychol Addict Behav. 2001 Dec;15(4):366-72. doi: 10.1037//0893-164x.15.4.366. PMID 11767270
- [Background] Weinstock H, Berman S, Cates W Jr. Sexually transmitted diseases among American youth: incidence and prevalence estimates, 2000. Perspect Sex Reprod Health. 2004 Jan-Feb;36(1):6-10. doi: 10.1363/psrh.36.6.04. PMID 14982671
- [Background] Winston FK, Mirman JH, Curry AE, Pfeiffer MR, Elliott MR, Durbin DR. Engagement with the TeenDrivingPlan and diversity of teens' supervised practice driving: lessons for internet-based learner driver interventions. Inj Prev. 2015 Feb;21(1):4-9. doi: 10.1136/injuryprev-2014-041212. Epub 2014 Jun 10. PMID 24916684
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Derived] Ford CA, Mirman JH, Garcia-Espana JF, Fisher Thiel MC, Friedrich E, Salek EC, Jaccard J. Effect of Primary Care Parent-Targeted Interventions on Parent-Adolescent Communication About Sexual Behavior and Alcohol Use: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199535. doi: 10.1001/jamanetworkopen.2019.9535. PMID 31418808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents between 14 and 17 years of age with an upcoming well-child visit and a parent were recruited from January 2016 through September 2016 from one urban primary care practice in the Pediatrics Research Consortium (PeRC) at Children's Hospital of Philadelphia (CHOP).
Pre-assignment Details: A total of 425 parent-adolescent dyads were contacted and screened. Of these, 188 (44%) did not meet eligibility criteria, 26 (6%) declined, and 37 (9%) could not be scheduled or reached again. 174 participant dyads we randomized into one of the five assignment groups.
Groups:
- Sexual Health (Teen): Teens between the ages of 14 and 15 will review psychoeducational workbooks related to sexual health at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Sexual Health: Psychoeducational workbook, worksheets, tip sheets, and health coaching session about sexual health, sexually transmitted disease (STD) prevention, and safe sex practices for teenager.
- Sexual Health (Parent): Parents of teens between the ages of 14 and 15 will review psychoeducational workbooks related to sexual health at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Sexual Health: Psychoeducational workbook, worksheets, tip sheets, and health coaching session about sexual health, sexually transmitted disease (STD) prevention, and safe sex practices for teenager.
- Alcohol Prevention (Teen): Teens between the ages of 14 and 15 will review psychoeducational workbooks related to alcohol prevention at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Alcohol Prevention: Psychoeducational workbook, worksheets, tip sheets, and health coaching session about alcohol prevention and safety, underage drinking, and drinking and driving.
- Alcohol Prevention (Parent): Parents of teens between the ages of 14 and 15 will review psychoeducational workbooks related to alcohol prevention at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Alcohol Prevention: Psychoeducational workbook, worksheets, tip sheets, and health coaching session about alcohol prevention and safety, underage drinking, and drinking and driving.
- Sexual Health & Alcohol Control Group (Teen): Teens between the ages of 14 and 15 will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 4 to 5 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from both the sexual health and alcohol prevention groups.
- Sexual Health & Alcohol Group (Parent): Parents of teens between the ages of 14 and 15 will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 4 to 5 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from both the sexual health and alcohol prevention groups.
- Teen Driving (Teen): Teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will review psychoeducational workbooks related to teen driving at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 6 months post baseline we will collect data to assess the effectiveness of the study materials.
  Teen Driving: Psychoeducational workbook, worksheets, videos, tip sheets, and health coaching session about how parents can help supervise their teens' safe driving practices and how to talk with their teen about important safety topics for teen drivers.
- Teen Driving (Parent): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will review psychoeducational workbooks related to teen driving at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 6 months post baseline we will collect data to assess the effectiveness of the study materials.
  Teen Driving: Psychoeducational workbook, worksheets, videos, tip sheets, and health coaching session about how parents can help supervise their teens' safe driving practices and how to talk with their teen about important safety topics for teen drivers.
- Teen Driving Control (Teen): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.
- Teen Driving Control (Parent): Teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.
Period: Overall Study
Arm/Group | Sexual Health (Teen) | Sexual Health (Parent) | Alcohol Prevention (Teen) | Alcohol Prevention (Parent) | Sexual Health & Alcohol Control Group (Teen) | Sexual Health & Alcohol Group (Parent) | Teen Driving (Teen) | Teen Driving (Parent) | Teen Driving Control (Teen) | Teen Driving Control (Parent)
Started | 40 | 40 | 40 | 40 | 40 | 40 | 28 | 28 | 26 | 26
Completed | 25 | 28 | 36 | 37 | 38 | 39 | 22 | 22 | 24 | 24
Not Completed | 15 | 12 | 4 | 3 | 2 | 1 | 6 | 6 | 2 | 2
Not completed — Lost to Follow-up | 11 | 9 | 4 | 3 | 2 | 1 | 6 | 6 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One sexual health dyad (2 participants) never completed Baseline so was withdrawn by PI. Another sexual health dyad (2 participants) was withdrawn by PI after the teen had difficulty completing study procedures due to cognitive delays.
Groups:
- Sexual Health & Alcohol Control Group (Parent): Parents of teens between the ages of 14 and 15 will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 4 to 5 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from both the sexual health and alcohol prevention groups.
- Teen Driving Control (Teens): Teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.
- Teen Driving Control (Parent): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.
- Total: Total of all reporting groups
Arm/Group | Sexual Health (Teen) | Sexual Health (Parent) | Alcohol Prevention (Teen) | Alcohol Prevention (Parent) | Sexual Health & Alcohol Control Group (Teen) | Sexual Health & Alcohol Control Group (Parent) | Teen Driving (Teen) | Teen Driving (Parent) | Teen Driving Control (Teens) | Teen Driving Control (Parent) | Total
Number analyzed (Participants) | 38 | 38 | 40 | 40 | 40 | 40 | 28 | 28 | 26 | 26 | 344
Age, Categorical [Count of Participants; unit: Participants] — Baseline characteristics were collected via survey.
  Participants
    <=18 years | 38 | 0 | 40 | 0 | 40 | 0 | 28 | 0 | 26 | 0 | 172
    Between 18 and 65 years | 0 | 37 | 0 | 40 | 0 | 40 | 0 | 28 | 0 | 25 | 170
    >=65 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.71 (.53) | 45.13 (8.6) | 14.83 (.53) | 45.20 (5.8) | 15.05 (.58) | 47.05 (5.9) | 16.81 (.56) | 46.57 (7.88) | 16.40 (.40) | 49.58 (8.50) | 31.13 (16.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 35 | 21 | 39 | 21 | 38 | 14 | 28 | 13 | 23 | 250
  Male | 20 | 3 | 19 | 1 | 19 | 2 | 14 | 0 | 13 | 3 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Asian | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 20 | 22 | 22 | 19 | 20 | 24 | 19 | 18 | 17 | 200
  White | 16 | 17 | 13 | 15 | 18 | 18 | 4 | 4 | 7 | 6 | 118
  More than one race | 2 | 1 | 2 | 3 | 1 | 1 | 0 | 4 | 1 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 38 | 40 | 40 | 40 | 40 | 28 | 28 | 26 | 26 | 344

OUTCOME MEASURES:

1. Primary Outcome: Quality of Parent-teen Communication (General- All Groups)
Description: Parents completed the 20-item Parent-Adolescent Communication Scale (PACS) (Barnes & Olson, 1985) which is scored such that a higher total score (sum of all items across scales) indicated better parent-adolescent communication. Teens answered the same questions, with only minor changes in wording when necessary. Scores were summed into an index that ranged from 41-96, α parent = 0.84, and 43-96, α teen = 0.87.
Time Frame: 4-6 months post-enrollment
Population: Arm 1 only. Parents and teens analyzed separately. Arm 2 (teen driving) had different primary outcomes (see outcomes 4-15) and therefore was not included here.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Alcohol (Teen): Parents of teens between the ages of 14 and 15 will review psychoeducational workbooks related to alcohol prevention at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 4 to 5 months post baseline we will collect data to assess the efficacy of the study materials.
  Alcohol Prevention: Psychoeducational workbook, worksheets, tip sheets, and health coaching session about alcohol prevention and safety, underage drinking, and drinking and driving.
- Sexual Health and Alcohol Control Group (Teen): Parents of teens between the ages of 14 and 15 will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 4 to 5 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from both the sexual health and alcohol prevention groups.
Arm/Group | Sexual Health (Parent) | Sexual Health (Teen) | Alcohol Prevention (Parent) | Alcohol (Teen) | Sexual Health & Alcohol Control Group (Parent) | Sexual Health and Alcohol Control Group (Teen)
Number analyzed (Participants) | 28 | 25 | 37 | 36 | 39 | 38
units on a scale | 77.8 (10.5) | 73.0 (9.4) | 77.2 (8.6) | 69.1 (8.4) | 77.4 (10.3) | 68.6 (11.1)
Statistical Analysis 1: Comparison: Alcohol Prevention (Parent) vs Sexual Health & Alcohol Control Group (Parent); Test type: Superiority; p = .906, Generalized Linear Model
Statistical Analysis 2: Comparison: Alcohol (Teen) vs Sexual Health and Alcohol Control Group (Teen); Test type: Superiority; p = .796, Generalized Linear Model
Statistical Analysis 3: Comparison: Sexual Health (Parent) vs Sexual Health & Alcohol Control Group (Parent); Test type: Superiority; p = .886, Generalized Linear Model
Statistical Analysis 4: Comparison: Sexual Health (Teen) vs Sexual Health and Alcohol Control Group (Teen); Test type: Other; p = .082, Generalized Linear Model

2. Primary Outcome: Frequency of Communication About Alcohol
Description: Frequency of communication about alcohol was measured with a single item followed by 4-point Likert-type response categories. Parents were asked: Since your teen's last well-child visit how much have you talked with your teen about alcohol? (Not at all (1), A little bit (2), Quite a bit (3), or A lot (4)). Teens were asked: Since your last well-child visit, how often have you and your (mother/father) talked about alcohol? (Never (1), Rarely (2), Sometimes (3), or Often (4)).
Time Frame: 4-6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sexual Health (Teen) | Sexual Health (Parent) | Alcohol Prevention (Teen) | Alcohol Prevention (Parent) | Sexual Health & Alcohol Control Group (Teen) | Sexual Health & Alcohol Group (Parent)
Number analyzed (Participants) | 25 | 28 | 36 | 37 | 38 | 39
units on a scale | 2.7 (1.0) | 2.5 (0.8) | 2.9 (0.8) | 2.6 (0.8) | 2.4 (1.2) | 2.5 (0.9)
Statistical Analysis 1: Comparison: Alcohol Prevention (Parent) vs Sexual Health & Alcohol Group (Parent); Test type: Superiority; p = 0.677, Generalized Linear Model
Statistical Analysis 2: Comparison: Alcohol Prevention (Teen) vs Sexual Health & Alcohol Control Group (Teen); Test type: Superiority; p = 0.020, Generalized Linear Model
Statistical Analysis 3: Comparison: Sexual Health (Parent) vs Sexual Health & Alcohol Group (Parent); Test type: Superiority; p = .952, Generalized Linear Model
Statistical Analysis 4: Comparison: Sexual Health (Teen) vs Sexual Health & Alcohol Group (Parent); Test type: Superiority; p = 0.210, Generalized Linear Model

3. Primary Outcome: Frequency of Communication About Sex
Description: Frequency of communication about sex was measured with a single item followed by 4-point Likert-type response categories. Parents were asked: Since your teen's last well-child visit how much have you talked with your teen about sex? (Not at all (1), A little bit (2), Quite a bit (3), or A lot (4)). Teens were asked: Since your last well-child visit, how often have you and your (mother/father) talked about sex? (Never (1), Rarely (2), Sometimes (3), or Often (4)).
Time Frame: 4-6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sexual Health (Teen) | Sexual Health (Parent) | Alcohol Prevention (Teen) | Alcohol Prevention (Parent) | Sexual Health & Alcohol Control Group (Teen) | Sexual Health & Alcohol Group (Parent)
Number analyzed (Participants) | 25 | 28 | 36 | 37 | 38 | 39
units on a scale | 2.3 (0.8) | 2.8 (0.8) | 2.1 (1.1) | 2.3 (0.9) | 1.8 (0.8) | 2.4 (1.0)
Statistical Analysis 1: Comparison: Alcohol Prevention (Parent) vs Sexual Health & Alcohol Group (Parent); Test type: Superiority; p = 0.505, Generalized Linear Model
Statistical Analysis 2: Comparison: Alcohol Prevention (Teen) vs Sexual Health & Alcohol Control Group (Teen); Test type: Superiority; p = .176, Generalized Linear Model
Statistical Analysis 3: Comparison: Sexual Health (Parent) vs Sexual Health & Alcohol Group (Parent); Test type: Superiority; p = 0.134, Generalized Linear Model
Statistical Analysis 4: Comparison: Sexual Health (Teen) vs Sexual Health & Alcohol Control Group (Teen); Test type: Superiority; p = 0.029, Generalized Linear Model

4. Primary Outcome: Parent-teen Communication About Reasons the Teen Wants to Drive
Description: Six months after baseline, parents reported on the frequency that they talked about reasons the teen wants to drive. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Teen Driving (Parents): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will review psychoeducational workbooks related to teen driving at a well-child visit appointment with the primary care giver (baseline); 2 weeks after baseline they will received a follow-up phone call and health coaching session to review the materials and ask questions; and then at 6 months post baseline we will collect data to assess the effectiveness of the study materials.
  Teen Driving: Psychoeducational workbook, worksheets, videos, tip sheets, and health coaching session about how parents can help supervise their teens' safe driving practices and how to talk with their teen about important safety topics for teen drivers.
- Teen Driving Control (Parents): Parents of teens between the ages of 16 and 17 who are planning on having the medical certification for the permit application completed and plan on taking their driving permit test in the next 8 weeks will receive their usual care at their well-child visit appointment with their primary care giver (baseline) and then at 6 months post baseline we will collect data. At the end of the post data collection, the control group will get all of the study materials from the teen driving group.
Arm/Group | Teen Driving (Parents) | Teen Driving Control (Parents)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.32 (.89) | 1.75 (.90)
Statistical Analysis 1: Comparison: Teen Driving (Parents) vs Teen Driving Control (Parents); Test type: Superiority; p = .037, t-test, 2 sided

5. Primary Outcome: Parent-teen Communication About the Kinds of Risky Driving Situations That Might Come up in His or Her Friend Group
Description: Six months after baseline, parents reported on the frequency that they talked about the kinds of risky driving situations that might come up in his or her friend group. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parents) | Teen Driving Control (Parents)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.59 (.73) | 1.79 (.98)
Statistical Analysis 1: Comparison: Teen Driving (Parents) vs Teen Driving Control (Parents); Test type: Superiority; p = .003, t-test, 2 sided

6. Primary Outcome: Parent-teen Communication About Pennsylvania's Graduated Driver Licensing Laws
Description: Six months after baseline, parents reported on the frequency that they talked about about Pennsylvania's GDL laws. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parents) | Teen Driving Control (Parents)
Number analyzed (Participants) | 22 | 24
units on a scale | 1.82 (.85) | .71 (1.08)
Statistical Analysis 1: Comparison: Teen Driving (Parents) vs Teen Driving Control (Parents); Test type: Superiority; p < .001, t-test, 2 sided

7. Primary Outcome: Parent-teen Communication About Wearing a Seatbelt
Description: Six months after baseline, parents reported on the frequency that they talked about wearing a seatbelt. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parents) | Teen Driving Control (Parents)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.68 (.72) | 2.79 (.59)
Statistical Analysis 1: Comparison: Teen Driving (Parents) vs Teen Driving Control (Parents); Test type: Superiority; p = .571, t-test, 2 sided

8. Primary Outcome: Parent-teen Communication About Dangers of Distracted Driving
Description: Six months after baseline, parents reported on the frequency that they talked about dangers of distracted driving. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parents) | Teen Driving Control (Parents)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.77 (.43) | 2.63 (.71)
Statistical Analysis 1: Comparison: Teen Driving (Parents) vs Teen Driving Control (Parents); Test type: Superiority; p = .394, t-test, 2 sided

9. Primary Outcome: Parent-teen Communication About Being a Safe Passenger
Description: Six months after baseline, parents reported on the frequency that they talked about being a safe passenger. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.55 (.67) | 1.71 (1.27)
Statistical Analysis 1: Comparison: Teen Driving (Parent) vs Teen Driving Control (Parent); Test type: Superiority; p = .008, t-test, 2 sided

10. Primary Outcome: Parent-teen Communication About What to do in a Crash
Description: Six months after baseline, parents reported on the frequency that they talked about what to do in a crash. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving | Teen Driving Control
Number analyzed (Participants) | 22 | 24
units on a scale | 2.00 (1.23) | .46 (.83)
Statistical Analysis 1: Comparison: Teen Driving vs Teen Driving Control; Test type: Superiority; p < .001, t-test, 2 sided

11. Primary Outcome: Parent-teen Communication About What to do if Stopped by a Police Officer
Description: Six months after baseline, parents reported on the frequency that they talked about what to do if stopped by a police officer. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.27 (.88) | 1.25 (1.07)
Statistical Analysis 1: Comparison: Teen Driving (Parent) vs Teen Driving Control (Parent); Test type: Superiority; p = .001, t-test, 2 sided

12. Primary Outcome: Parent-teen Communication About Driving Under the Influence of Drugs or Alcohol
Description: Six months after baseline, parents reported on the frequency that they talked about driving under the influence of drugs or alcohol. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 1.73 (1.16) | 1.21 (1.29)
Statistical Analysis 1: Comparison: Teen Driving (Parent) vs Teen Driving Control (Parent); Test type: Superiority; p = .159, t-test, 2 sided

13. Primary Outcome: Parent-teen Communication About What to do if the Teen Needs a Safe Ride Home
Description: Six months after baseline, parents reported on the frequency that they talked about what to do if the teen needs a safe ride home. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.45 (.86) | 1.96 (1.20)
Statistical Analysis 1: Comparison: Teen Driving (Parent) vs Teen Driving Control (Parent); Test type: Superiority; p = .112, t-test, 2 sided

14. Primary Outcome: Parent-teen Communication About Stopping a Friend From Driving Under the Influence of Drugs or Alcohol
Description: Six months after baseline, parents reported on the frequency that they talked about stopping a friend from driving under the influence of drugs or alcohol. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).stopping a friend from riding with a driver who is under the influence of drugs or alcohol
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 2.64 (.66) | 2.29 (.955)
Statistical Analysis 1: Comparison: Teen Driving (Parent); Test type: Superiority; p = .165, t-test, 2 sided

15. Primary Outcome: Parent-teen Communication About Stopping a Friend From Riding With a Driver Who is Under the Influence of Drugs or Alcohol
Description: Six months after baseline, parents reported on the frequency that they talked about stopping a friend from riding with a driver who is under the influence of drugs or alcohol. Parents selected from one of the following response choices: "never talked about" (0); "talked about once or twice" (1); "talked about three or four times" (2); "talked about a lot, about 5 times or more" (3).
Time Frame: 6 months post-enrollment
Population: Parent Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teen Driving (Parent) | Teen Driving Control (Parent)
Number analyzed (Participants) | 22 | 24
units on a scale | 1.68 (1.17) | .71 (1.12)
Statistical Analysis 1: Comparison: Teen Driving (Parent) vs Teen Driving Control (Parent); Test type: Superiority; p = .006, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each time point (e.g. Baseline, 2wk follow up, final follow up).
Arm/Group | Sexual Health | Alcohol Prevention | Sexual Health & Alcohol Control Group | Teen Driving | Teen Driving Control
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/56 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/56 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT02554682/Prot_SAP_000.pdf